CLINICAL TRIAL: NCT01946776
Title: Cardiac Arrhythmias in Refractory Epilepsy: Identifying Prevalence and LINKage Between Seizures and Arrhythmias
Brief Title: Cardiac Arrhythmias in Epilepsy: the CARELINK-study
Acronym: CARELINK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stichting Epilepsie Instellingen Nederland (Other)
Collaborators: Fonds NutsOhra (Other); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1201-071
Record Dates: First submitted 2013-08-29; First posted 2013-09-20 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Epilepsy; Asystole; Cardiac Arrhythmias
MeSH Terms: conditions — Epilepsy; Heart Arrest; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reveal XT (Other): People with drug-resistant epilepsy whose heart rhythm will be monitored continuously for 2 years using Reveal XT, an implantable heart rate monitor.
  Interventions: Device: implantable heart rate monitor

INTERVENTIONS:
Device: implantable heart rate monitor — Implantation of Reveal XT
  Other Names: Reveal XT

SUMMARY:
Patients with difficult-to-treat epilepsy ("refractory epilepsy") are at high risk of sudden death: sudden unexpected death in epilepsy (SUDEP). Cardiac arrhythmias are one of the possible causes of SUDEP. When monitoring in the hospital setting, the frequency of cardiac arrhythmias in people with epilepsy is low: 0,4%. However, when a subcutaneous implantable device (Reveal XT) is used to monitor heart rhythm continuously for an extended period of time, the frequency of clinically relevant arrhythmias appeared much higher in two small observational studies (n=19): 6-20%. The aim of this study is to analyze the frequency and underlying mechanism of cardiac arrhythmias in a larger group of 50 people with refractory epilepsy with Reveal XT. In the future, this may help us to identify those epilepsy patients at high risk of cardiac arrhythmias, so that we can timely institute preventive measures (e.g. pacemaker implantation).

ELIGIBILITY:
Inclusion Criteria:

* Drug-resistant focal epilepsy: failure of adequate trials of two tolerated and appropriately chosen and used antiepileptic drug (AED) schedules (whether as monotherapies or in combination) to achieve sustained seizure freedom [16]
* ≥ 1 complex partial and/or generalized tonic clonic seizure/month as indicated by history taking
* If female, not pregnant
* Aged 18 to 60 years
* Able to undergo the study procedure as judged by the treating physician.

Exclusion Criteria:

* Clinical suspicion of seizure-induced asystole (e.g. seizures with sudden flaccid falls)
* Reveal implantation (either present or in the past)
* Known clinical relevant structural cardiac disease
* Hereditary syndromes that increase the risk of cardiomyopathy (e.g. Marfan's disease)
* ECG findings suggestive of arrhythmias without proper cardiac evaluation to in- or exclude this possibility. According to European Society of Cardiology (ESC) guidelines on syncope the following ECG findings will be used: bifascicular block and other intraventricular conduction abnormalities, asymptomatic inappropriate sinus bradycardia (<50 bpm), sinoatrial block or sinus pause ≥3s in the absence of negative chronotropic medications, non-sustained VT, pre-exited QRS complexes, prolonged or short QT interval, Brugada pattern, pattern suggestive of arrhythmogenic right ventricular cardiomyopathy.
* Pacemaker
* Use of beta blockers or other anti-arrhythmic/anti-arrhythmogenic medication
* Previous diagnosis of psychogenic non-epileptic seizures
* Patients who live alone and are not able to recall their seizures

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence and two-year prevalence of clinically relevant cardiac arrhythmia. | Continuously for two years or until the end-of-battery-life of Reveal XT (this period is expected to last an additional six months on average)
  Clinical relevant cardiac arrhythmia is defined as:
  1. Asystole of ≥ 6s together with clinical symptoms (lightheadedness, syncope, seizure) as indicated by seizure diary, activation of the portable seizure monitor, or patient activation of Reveal XT. The time frame between the reported clinical symptoms and the recorded event should not exceed 15 minutes.
  2. Asystole of ≥10s regardless of report of clinical symptoms
  3. Other cardiac arrhythmias of clinical significance:
     1. polymorphic sustained or non-sustained ventricular tachycardia (VT)
     2. non-sustained monomorphic VT of >180 bpm and >2s duration, or >175 bpm and >3s duration, and sustained monomorphic VT
     3. atrial fibrillation (AF) of >200 bpm and >30s duration, or <55 bpm and clinical symptoms (dizziness or dyspnea)
     4. persistent sinus bradycardia of <40 bpm during physical activity
     5. asymptomatic 2nd or 3rd degree atrioventricular (AV) block of >4s duration

SECONDARY OUTCOMES:
the number of patients who will have received a permanent pacemaker at the end of this study. | Continuously for two years or until the end-of-battery-life of Reveal XT (this period is expected to last an additional six months on average)
  Participants who will exhibit a clinically relevant arrhythmia (see our primary endpoints) during this study will be referred to an independent cardiologist for further evaluation and/or treatment. In a certain number of cases, this cardiologist will decide with the patient that pacemaker implantation would be the appropriate cause of action.

OTHER OUTCOMES:
The percentage of seizure-related cardiac arrhythmias | Continuously for two years or until the end-of-battery-life of Reveal XT (this period is expected to last an additional six months on average)
  The number of seizures during which a cardiac arrhythmia occurs divided by the total number of seizures during this study
The percentage of patients with a cardioinhibitory response to head-up tilt-testing | During one head-up tilt-test (approximate duration 1,5 hours)
  The number of patients with a cardioinhibitory response to head-up tilt-testing (1) heart rate rising initially then falling to a ventricular rate of <40 bpm for >10 seconds or asystole occurring for >3 seconds, with blood pressure rising initially then falling before the heart rate falls 2) Heart rate rising initially then falling to a ventricular rate <40 bpm for >10 seconds or asystole occurring for >3 seconds, with blood pressure rising initially and only falling to hypotensive levels <80 mm Hg systolic at or after the onset of rapid and severe heart rate fall) divided by the number of patients in whom tilt-testing was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Roland D Thijs, PhD, Principal Investigator — SEIN-Epilepsy Institute in the Netherlands Foundation
Locations (4):
- Netherlands (4):
  - Atrium Medical Center, Heerlen
  - Epilepsy center Kempenhaeghe, Heeze
  - Epilepsy Instititute in the Netherlands Foundation (SEIN), Hoofddorp
  - Antonius Hospital, Sneek

REFERENCES:
- [Background] Surges R, Thijs RD, Tan HL, Sander JW. Sudden unexpected death in epilepsy: risk factors and potential pathomechanisms. Nat Rev Neurol. 2009 Sep;5(9):492-504. doi: 10.1038/nrneurol.2009.118. Epub 2009 Aug 11. PMID 19668244
- [Background] Schuele SU, Bermeo AC, Alexopoulos AV, Locatelli ER, Burgess RC, Dinner DS, Foldvary-Schaefer N. Video-electrographic and clinical features in patients with ictal asystole. Neurology. 2007 Jul 31;69(5):434-41. doi: 10.1212/01.wnl.0000266595.77885.7f. PMID 17664402
- [Background] Rugg-Gunn FJ, Simister RJ, Squirrell M, Holdright DR, Duncan JS. Cardiac arrhythmias in focal epilepsy: a prospective long-term study. Lancet. 2004 Dec 18-31;364(9452):2212-9. doi: 10.1016/S0140-6736(04)17594-6. PMID 15610808
- [Background] Nei M, Sperling MR, Mintzer S, Ho RT. Long-term cardiac rhythm and repolarization abnormalities in refractory focal and generalized epilepsy. Epilepsia. 2012 Aug;53(8):e137-40. doi: 10.1111/j.1528-1167.2012.03561.x. Epub 2012 Jun 18. PMID 22709423
- [Background] Sevcencu C, Struijk JJ. Autonomic alterations and cardiac changes in epilepsy. Epilepsia. 2010 May;51(5):725-37. doi: 10.1111/j.1528-1167.2009.02479.x. Epub 2010 Jan 7. PMID 20067509